CLINICAL TRIAL: NCT00865709
Title: Phase 2b, DB, Randomized Study Evaluating Efficacy & Safety of Sorafenib Compared With Placebo When Administered in Combination With Modified FOLFOX6 for the Treatment of Metastatic CRC Subjects Previously Untreated for Stage IV Disease
Brief Title: Study of Modified FOLFOX6 Plus or Minus Sorafenib in Stage IV Metastatic Colorectal Carcinoma (mCRC) Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13162; 2008-005025-11 (EudraCT Number)
Record Dates: First submitted 2009-02-02; First posted 2009-03-19 (Estimated); Results first posted 2012-03-20 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-11

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Colorectal Cancer; Metastasis; Stage IV; Liver Metastasis
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — Sorafenib; Fluorouracil; Levoleucovorin; Oxaliplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sorafenib (Nexavar, BAY43-9006) + mFOLFOX6 (Experimental): Subjects will receive oral Sorafenib 400 mg twice daily (BID) continuously and intravenous (IV) mFOLFOX6 (5-FU 400 mg/m^2 bolus and 2400 mg/m^2 for 46-48 hrs; levo-leucovorin 200 mg/m^2; 85 mg/m^2 oxaliplatin) every 14 days until progressive disease (PD)
  Interventions: Drug: Sorafenib (Nexavar, BAY43-9006) + mFOLFOX6 (5-FU, levo-leucovorin, oxaliplatin)
- Matching placebo + mFOLFOX6 (Placebo Comparator): Subjects will receive oral matching placebo 2 tablets BID continuously and IV mFOLFOX6 (5-FU 400 mg/m^2 bolus and 2400 mg/m^2 for 46-48 hrs; levo-leucovorin 200 mg/m^2; 85 mg/m^2 oxaliplatin) every 14 days until progressive disease
  Interventions: Drug: Matching placebo + mFOLFOX6 (5-FU, levo-leucovorin, oxaliplatin)

INTERVENTIONS:
Drug: Sorafenib (Nexavar, BAY43-9006) + mFOLFOX6 (5-FU, levo-leucovorin, oxaliplatin) — Subjects will receive oral Sorafenib 400 mg twice daily (BID) continuously and intravenous (IV) mFOLFOX6 (5-FU 400 mg/m^2 bolus and 2400 mg/m^2 for 46-48 hrs; levo-leucovorin 200 mg/m^2; 85 mg/m^2 oxaliplatin) every 14 days until progressive disease (PD)
  Arms: Sorafenib (Nexavar, BAY43-9006) + mFOLFOX6
Drug: Matching placebo + mFOLFOX6 (5-FU, levo-leucovorin, oxaliplatin) — Subjects will receive oral matching placebo 2 tablets BID continuously and IV mFOLFOX6 (5-FU 400 mg/m^2 bolus and 2400 mg/m^2 for 46-48 hrs; levo-leucovorin 200 mg/m^2; 85 mg/m^2 oxaliplatin) every 14 days until progressive disease
  Arms: Matching placebo + mFOLFOX6

SUMMARY:
To determine if sorafenib when added to chemotherapy will slow disease progression more than chemotherapy alone in patients previously untreated for metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of adenocarcinoma of the colon or rectum
* Tumor tissue sample available for KRAS and BRAF assessment
* Measurable metastatic Stage IV disease including at least one measurable lesion that has not previously been radiated
* No prior chemotherapy for metastatic CRC
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1
* Life expectancy of at least 12 weeks
* Adequate bone marrow, liver, and renal function; adequate clotting parameters

Exclusion Criteria:

* Prior treatment with sorafenib
* Clinical or radiographic evidence of brain metastasis
* Major surgery, surgical biopsy, or significant traumatic injury within 28 days of randomization; evidence or history of bleeding diathesis or coagulopathy
* Red blood cell (RBC), white blood cell (WBC), or platelet transfusions and/or growth factor use within 28 days before randomization
* Adjuvant therapy for CRC (Stage I, II, or III) completed within 12 months before randomization
* Serious, non-healing wound, ulcer, or bone fracture; Grade 3 or 4 hemorrhage within 28 days before randomization
* Use of anticoagulation therapy (low dose anticoagulation therapy to mitigate risk of thrombosis due to placement of a semi-permanent central venous port for administration of chemotherapy is allowed. The use of coumadin and related compounds is excluded.)
* Uncontrolled hypertension (systolic blood pressure > 150 mmHg or diastolic pressure > 100 mmHg on repeated measurement) despite optimal medical management
* Thrombolic, embolic, venous, or arterial events (eg, cerebrovascular accident, including transient ischemic attacks) within 6 months before randomization
* Active cardiac disease including:

  * Congestive heart failure
  * Unstable angina or myocardial infarction within the 6 months before randomization
  * Cardiac ventricular arrhythmias requiring antiarrhythmic treatment
* Peripheral neuropathy > Grade 1 (CTCAE)
* Known HIV infection or chronic hepatitis B or C infection
* Any active infection >/= Grade 2 (CTCAE)
* Any medical, psychological, or social condition that may interfere with the subject's participation in the study or evaluation of the study results
* Use of any investigational drug within 28 days or 5 half-lives of that drug, whichever is longer, before randomization
* Subjects with metastatic CRC who are currently candidates for surgery with curative intent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2009-03; Primary Completion 2011-01 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (102):
- United States (5):
  - Wichita, Kansas
  - Metairie, Louisiana
  - Brockton, Massachusetts
  - Burlington, Massachusetts
  - Dallas, Texas
- Belgium (5):
  - Antwerp
  - Bruxelles - Brussel
  - Ghent
  - Leuven
  - Liège
- Hungary (6):
  - Budapest
  - Debrecen
  - Győr
  - Kecskemét
  - Szeged
  - Székesfehérvár
- Italy (8):
  - Castelfranco Veneto, Treviso
  - Genova
  - Macerata
  - Palermo
  - Pordenone
  - Torino
  - Udine
  - Verona
- Poland (8):
  - Bialystok
  - Elblag
  - Gdansk
  - Gdynia
  - Krakow
  - Olsztyn
  - Warsaw
  - Wroclaw
- Romania (9):
  - Alba Iulia
  - Baia Mare
  - Bucharest
  - Cluj-Napoca
  - Craiova-Dolj
  - Iași
  - Oradea
  - Suceava
  - Timișoara
- Russia (27):
  - Arkhangelsk
  - Astrakhan
  - Chelyabinsk
  - Irkutsk
  - Ivanovo
  - Izhevsk
  - Kazan'
  - Khabarovsk
  - Krasnodar
  - Kursk
  - Magnitogorsk
  - Moscow
  - Nizhny Novgorod
  - Novosibirsk
  - Obninsk
  - Pjatygorsk
  - Rostov-on-Don
  - Saint Petersburg
  - Samara
  - Sochi
  - Syktyvkar
  - Tula
  - Ulyanovsk
  - Vladimir
  - Volgograd
  - Yaroslavl
  - Yekaterinburg
- Spain (9):
  - Barcelona, Barcelona
  - L'Hospitalet de Llobregat, Barcelona
  - Manresa, Barcelona
  - Santander, Cantabria
  - Palma de Mallorca, Illes Baleares
  - Málaga, Málaga
  - Seville, Sevilla
  - Valencia, Valencia
  - Madrid
- Ukraine (13):
  - Cherkassy
  - Dnipro
  - Dnipropetrovsk
  - Donetsk
  - Ivano-Frankivsk
  - Kharkiv
  - Kiev
  - Kryvyi Rih
  - Luhansk
  - Lviv
  - Mariupol
  - Sumy
  - Uzhhorod
- United Kingdom (12):
  - Bristol, Avon
  - Manchester, Manchester
  - Liverpool, Merseyside
  - Northwood, Middlesex
  - Nottingham, Nottinghamshire
  - Aberdeen
  - Belfast
  - Glasgow
  - Hull
  - London
  - Newcastle upon Tyne
  - Portsmouth

REFERENCES:
- [Result] Tabernero J, Garcia-Carbonero R, Cassidy J, Sobrero A, Van Cutsem E, Kohne CH, Tejpar S, Gladkov O, Davidenko I, Salazar R, Vladimirova L, Cheporov S, Burdaeva O, Rivera F, Samuel L, Bulavina I, Potter V, Chang YL, Lokker NA, O'Dwyer PJ. Sorafenib in combination with oxaliplatin, leucovorin, and fluorouracil (modified FOLFOX6) as first-line treatment of metastatic colorectal cancer: the RESPECT trial. Clin Cancer Res. 2013 May 1;19(9):2541-50. doi: 10.1158/1078-0432.CCR-13-0107. Epub 2013 Mar 26. PMID 23532888
- See also: Click here and search for Bayer Product information provided by the EMA — http://www.clinicaltrialsregister.eu

RESULTS

PARTICIPANT FLOW:
Period: Treatment
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + mFOLFOX6 | Matching Placebo + mFOLFOX6
Started | 97 | 101
Received Treatment | 97 (Safety population) | 101 (Safety population)
Completed | 67 (Patients who continued treatment at data cut-off or discontinued treatment due to PD or death) | 83 (Patients who continued treatment at data cut-off or discontinued treatment due to PD or death)
Not Completed | 30 | 18
Not completed — Adverse Event | 9 | 6
Not completed — Withdrawal by Subject | 10 | 7
Not completed — Physician Decision | 3 | 2
Not completed — Surgery | 8 | 3
Period: Active Follow-up
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + mFOLFOX6 | Matching Placebo + mFOLFOX6
Started | 25 | 16
Completed | 17 | 15
Not Completed | 8 | 1
Period: Long Term Follow-up
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + mFOLFOX6 | Matching Placebo + mFOLFOX6
Started | 70 | 82
Completed | 24 | 33
Not Completed | 46 | 49

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + mFOLFOX6 | Matching Placebo + mFOLFOX6 | Total
Number analyzed (Participants) | 97 | 101 | 198
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (10.3) | 60.3 (8.3) | 59.8 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 38 | 93
  Male | 42 | 63 | 105
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4
  Spain | 25 | 25 | 50
  Belgium | 1 | 0 | 1
  Romania | 3 | 8 | 11
  Russian Federation | 54 | 52 | 106
  United Kingdom | 12 | 14 | 26
ECOG (Eastern Cooperative Oncology Group) Performance Status [Number; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status is a scale that measures how cancer affects the daily life of a patient on an ordinal scale from grade 0 (best) to grade 5 (worst).
  Participants
    0=Fully active without restriction | 34 | 36 | 70
    1= Restricted in physically strenuous activity | 63 | 65 | 128
    2= Ambulatory, capable of all selfcare | 0 | 0 | 0
    3= Capable of limited selfcare | 0 | 0 | 0
    4= Completely disabled | 0 | 0 | 0
    5= Dead | 0 | 0 | 0
Stage of Disease at study entry (TNM Classification, Stage IV) [Number; unit: Participants] — The TNM (Tumor, Nodes, Metastasis) classification is a three-dimensional solid tumor classification system. The "T" dimension categorizes the size and degree of tumor spreading on an ordinal scale from T0 (best) to T4 (worst). The "N" dimension categorizes the degree of spreading of the tumor into lymph nodes on an ordinal scale from N0 (best) to N3 (worst). The "M" dimension categorizes whether or not the cancer has metastases beyond the lymph nodes on an ordinal scale from M0 (no metastases) to M1 (metastases). All of the 198 randomized patients were at Stage IV of disease.
  Participants | 97 | 101 | 198
Time since initial diagnosis [Mean (Standard Deviation); unit: Months] — Time since initial diagnosis was the mean time from initial diagnosis to randomization into the study.
  Months | 9.8 (16.2) | 9.2 (16.9) | 9.5 (16.6)
Liver metastases by Principal Investigator [Number; unit: Participants] — Liver metastases by Principal Investigator
  Participants
    Yes | 79 | 81 | 160
    No | 18 | 20 | 38
Number of metastatic sites by Principal Investigator [Number; unit: Participants] — Number of metastatic sites by Principal Investigator
  Participants
    <3 | 71 | 71 | 142
    >=3 | 26 | 30 | 56
KRAS [Number; unit: Participants] — Kirsten rat sarcoma viral oncogene homolog (KRAS)
  Participants
    Mutant | 33 | 43 | 76
    Wild-Type | 42 | 41 | 83
    Missing | 22 | 17 | 39

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: Progression-free Survival (PFS) was defined as the time from date of randomization to disease progression or death due to any cause, whichever occurred first. Subjects without progression or death at the time of analysis were censored at their last date of tumor evaluation. Disease progression was defined as an increase of at least 20% in the sum of tumor lesions sizes.
Time Frame: From randomization of the first subject until 23 months later, assessed every 8 weeks.
Population: The test was conducted using the intent-to-treat (ITT) population (all subjects who were randomized).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + mFOLFOX6 | Matching Placebo + mFOLFOX6
Number analyzed (Participants) | 97 | 101
Months | 9.1 [7.6 to 9.7] | 8.7 [7.4 to 9.5]
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) + mFOLFOX6 vs Matching Placebo + mFOLFOX6; A sample size of 120 PFS events would provide a > 85% power at a target HR = 0.65 between sorafenib and matching placebo, with a 1-sided alpha = 0.10, for testing the null hypothesis H0: HR ≥ 1 versus the alternative hypothesis H1: HR < 1 based on the log-rank test. The test was conducted using the intent-to-treat (ITT) population, defined as all subjects who were randomized to treatment; Test type: Superiority or Other; p = 0.2309, Log Rank — 1-sided p-value from stratified log-rank test, stratified by factors of # metastatic sites and liver metastasis determined by Principal Investigator; Hazard Ratio (HR) = 0.884, 95% CI 2-sided [0.635 to 1.231] — The relative risk (sorafenib to placebo) was estimated by the hazard ratio from stratified Cox regression with a 95% confidence interval

2. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) was defined as the time from date of randomization to death due to any cause. Subjects still alive at the time of analysis were censored at their last date of last contact.
Time Frame: From randomization of the first subject until 33 months later.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + mFOLFOX6 | Matching Placebo + mFOLFOX6
Number analyzed (Participants) | 97 | 101
days | 535 [437 to 613] | 552 [453 to 651]

3. Secondary Outcome: Time to Progression (TTP)
Description: Time to progression (TTP) was defined as the time from date of randomization to disease progression. Subjects without progression at the time of analysis were censored at their last date of tumor evaluation. Disease progression was defined as an increase of at least 20% in the sum of tumor lesions sizes.
Time Frame: From randomization of the first subject until 23 months later, assessed every 8 weeks.
Population: The test was conducted using the intent-to-treat (ITT) population (all subjects who were randomized).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + mFOLFOX6 | Matching Placebo + mFOLFOX6
Number analyzed (Participants) | 97 | 101
Months | 9.2 [7.8 to 11.0] | 9.0 [7.6 to 10.4]
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) + mFOLFOX6 vs Matching Placebo + mFOLFOX6; A sample size of 120 PDs would provide a > 85% power at a target HR = 0.65 between sorafenib and matching placebo, with a 1-sided alpha = 0.10, for testing H0: HR ≥ 1 versus H1: HR < 1 based on the log-rank test. The test was conducted using the intent-to-treat (ITT) population (all subjects who were randomized); Test type: Superiority or Other; p = 0.1437, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.829, 95% CI 2-sided [0.586 to 1.174] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Overall Response
Description: Overall response of a subject was defined as the best tumor response (Complete Response (CR) or Partial Response (PR)) observed during trial period assessed according to the Response Evaluation Criteria in Solid Tumors (RECIST) criteria. CR was defined as disappearance of tumor lesions, PR was defined as a decrease of at least 30% in the sum of tumor lesion sizes.
Time Frame: From randomization of the first subject until 23 months later, assessed every 8 weeks.
Population: The test was conducted using the intent-to-treat (ITT) population (all subjects who were randomized).
Measure: Number; unit: participants
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + mFOLFOX6 | Matching Placebo + mFOLFOX6
Number analyzed (Participants) | 97 | 101
participants | 45 | 61
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) + mFOLFOX6 vs Matching Placebo + mFOLFOX6; The proportion of subjects achieving overall response (CR or PR), when confirmation of response was not required, was estimated with a 95% confidence interval for each treatment group. The treatment groups were compared with respect to overall response rate using the Cochran-Mantel-Haenszel test, adjusting for the stratification factors; Test type: Superiority or Other; p = 0.023, Cochran-Mantel-Haenszel — 1-sided p-value from the Cochran-Mantel-Haenszel test, adjusting for the stratification factors of # metastatic sites and liver metastasis determined by Principal Investigator

5. Secondary Outcome: Duration of Response
Description: Duration of Response was defined as the time from date of first response (Complete Response (CR) or Partial Response (PR)) to the date when Progressive Disease (PD) was first documented or to the date of death, whichever occurred first according to Response Evaluation Criteria in Solid Tumors (RECIST). Subjects still having CR or PR and alive at the time of analysis were censored at their last date of tumor evaluation. CR was defined as disappearance of tumor lesions, PR as a decrease of at least 30% and PD as an increase of at least 20% in the sum of tumor lesions sizes.
Time Frame: From randomization of the first subject until 23 months later, assessed every 8 weeks
Population: Duration of response was the time from the first documented CR or PR until the first documented PD or death (if before progression). Only responders (CR or PR) were included in the analysis
Measure: Number (95% Confidence Interval); unit: months
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + mFOLFOX6 | Matching Placebo + mFOLFOX6
Number analyzed (Participants) | 45 | 61
months | 7.5 [5.7 to 9.4] | 6.7 [5.5 to 8.1]

ADVERSE EVENTS:
Time Frame: All adverse events from consent to 30 days after last dose of study drug. From randomization of first subject until 23 months later. From randomization of first subject until 33 months later (OS update).
Description: Other Adverse Events below includes all reported treatment emergent adverse events (total of all non-serious and serious adverse events) for the provided MedDRA Preferred Terms
Groups:
- Sorafenib (Nexavar, BAY43-9006) + mFOLFOX6 (OS Update): Subjects will receive oral Sorafenib 400 mg twice daily (BID) continuously and intravenous (IV) mFOLFOX6 (5-FU 400 mg/m^2 bolus and 2400 mg/m^2 for 46-48 hrs; levo-leucovorin 200 mg/m^2; 85 mg/m^2 oxaliplatin) every 14 days until progressive disease (PD)
- Matching Placebo + mFOLFOX6 (OS Update): Subjects will receive oral matching placebo 2 tablets BID continuously and IV mFOLFOX6 (5-FU 400 mg/m^2 bolus and 2400 mg/m^2 for 46-48 hrs; levo-leucovorin 200 mg/m^2; 85 mg/m^2 oxaliplatin) every 14 days until progressive disease
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + mFOLFOX6 | Matching Placebo + mFOLFOX6 | Sorafenib (Nexavar, BAY43-9006) + mFOLFOX6 (OS Update) | Matching Placebo + mFOLFOX6 (OS Update)
Serious Adverse Events (participants affected / at risk) | 30/97 | 27/101 | 33/97 | 30/101
Other Adverse Events (participants affected / at risk) | 96/97 | 99/101 | 96/97 | 99/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib (Nexavar, BAY43-9006) + mFOLFOX6 (N=97) | Matching Placebo + mFOLFOX6 (N=101) | Sorafenib (Nexavar, BAY43-9006) + mFOLFOX6 (OS Update) (N=97) | Matching Placebo + mFOLFOX6 (OS Update) (N=101)
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 2 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 3 | 0 | 5
Vomiting (Gastrointestinal disorders) | 1 | 2 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 1 | 2
Large intestine perforation (Gastrointestinal disorders) | 1 | 1 | 1 | 1
Subileus (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Colonic obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Duodenal perforation (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Enterovesical fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Device related infection (Infections and infestations) | 1 | 2 | 1 | 2
Cellulitis (Infections and infestations) | 1 | 1 | 1 | 1
Abdominal abscess (Infections and infestations) | 0 | 1 | 0 | 1
Diabetic foot infection (Infections and infestations) | 1 | 0 | 1 | 0
Gastroenteritis salmonella (Infections and infestations) | 0 | 1 | 0 | 1
Lobar pneumonia (Infections and infestations) | 0 | 1 | 0 | 1
Osteomyelitis (Infections and infestations) | 1 | 0 | 1 | 0
Peritoneal infection (Infections and infestations) | 0 | 1 | 0 | 1
Proctitis bacterial (Infections and infestations) | 1 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 1 | 1 | 1
Chest discomfort (General disorders) | 0 | 1 | 0 | 1
Device breakage (General disorders) | 1 | 0 | 1 | 0
Disease progression (General disorders) | 0 | 1 | 1 | 1
Mucosal inflammation (General disorders) | 1 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 1 | 1 | 1
Renal failure acute (Renal and urinary disorders) | 2 | 0 | 2 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 1
Cardiovascular insufficiency (Cardiac disorders) | 0 | 1 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 1
Axillary vein thrombosis (Vascular disorders) | 1 | 0 | 1 | 0
Circulatory collapse (Vascular disorders) | 1 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1 | 0 | 1
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 1 | 3
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0 | 1 | 0
Blood amylase increased (Investigations) | 0 | 1 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Retinal vein thrombosis (Eye disorders) | 1 | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0 | 1 | 0
Metasteses to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib (Nexavar, BAY43-9006) + mFOLFOX6 (N=97) | Matching Placebo + mFOLFOX6 (N=101) | Sorafenib (Nexavar, BAY43-9006) + mFOLFOX6 (OS Update) (N=97) | Matching Placebo + mFOLFOX6 (OS Update) (N=101)
Diarrhoea (Gastrointestinal disorders) | 49 | 39 | 49 | 39
Nausea (Gastrointestinal disorders) | 36 | 49 | 36 | 49
Vomiting (Gastrointestinal disorders) | 24 | 20 | 24 | 22
Abdominal pain (Gastrointestinal disorders) | 15 | 23 | 16 | 23
Constipation (Gastrointestinal disorders) | 12 | 21 | 12 | 21
Stomatitis (Gastrointestinal disorders) | 22 | 4 | 22 | 5
Abdominal pain upper (Gastrointestinal disorders) | 8 | 6 | 8 | 7
Dyspepsia (Gastrointestinal disorders) | 3 | 6 | 3 | 6
Rectal haemorrhage (Gastrointestinal disorders) | 5 | 4 | 5 | 3
Abdominal pain lower (Gastrointestinal disorders) | 2 | 5 | 2 | 5
Abdominal distension (Gastrointestinal disorders) | 1 | 5 | 1 | 7
Proctalgia (Gastrointestinal disorders) | 5 | 0 | 5 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 22 | 25 | 22 | 25
Dysaesthesia (Nervous system disorders) | 16 | 21 | 16 | 21
Neurotoxicity (Nervous system disorders) | 19 | 13 | 19 | 13
Paraesthesia (Nervous system disorders) | 10 | 20 | 10 | 19
Neuropathy peripheral (Nervous system disorders) | 13 | 9 | 13 | 10
Dysgeusia (Nervous system disorders) | 12 | 6 | 12 | 6
Hypoaesthesia (Nervous system disorders) | 9 | 9 | 9 | 9
Dizziness (Nervous system disorders) | 6 | 10 | 6 | 10
Headache (Nervous system disorders) | 6 | 3 | 6 | 4
Lethargy (Nervous system disorders) | 2 | 5 | 2 | 5
Asthenia (General disorders) | 31 | 24 | 31 | 24
Fatigue (General disorders) | 22 | 24 | 22 | 24
Mucosal inflammation (General disorders) | 21 | 16 | 21 | 16
Pyrexia (General disorders) | 10 | 11 | 10 | 11
Oedema peripheral (General disorders) | 3 | 6 | 3 | 6
Neutropenia (Blood and lymphatic system disorders) | 60 | 39 | 60 | 39
Thrombocytopenia (Blood and lymphatic system disorders) | 18 | 25 | 18 | 25
Anaemia (Blood and lymphatic system disorders) | 23 | 15 | 23 | 15
Leukopenia (Blood and lymphatic system disorders) | 11 | 7 | 11 | 7
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 52 | 11 | 52 | 11
Rash (Skin and subcutaneous tissue disorders) | 23 | 10 | 24 | 10
Alopecia (Skin and subcutaneous tissue disorders) | 23 | 6 | 23 | 6
Dry skin (Skin and subcutaneous tissue disorders) | 7 | 8 | 7 | 8
Erythema (Skin and subcutaneous tissue disorders) | 11 | 4 | 12 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 3 | 5 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 | 10 | 9 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 8 | 9 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 10 | 6 | 10
Dysaesthesia pharynx (Respiratory, thoracic and mediastinal disorders) | 3 | 6 | 3 | 6
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 | 6 | 2 | 6
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 2 | 5
Upper respiratory tract infection (Infections and infestations) | 0 | 5 | 0 | 5
Blood amylase increased (Investigations) | 5 | 10 | 5 | 10
Platelet count decreased (Investigations) | 3 | 8 | 3 | 8
Aspartate aminotransferase increased (Investigations) | 5 | 5 | 5 | 7
Lipase increased (Investigations) | 6 | 4 | 6 | 4
Alanine aminotransferase increased (Investigations) | 4 | 5 | 4 | 6
Weight decreased (Investigations) | 5 | 1 | 5 | 1
Neutrophil count decreased (Investigations) | 0 | 5 | 0 | 5
Decreased appetite (Metabolism and nutrition disorders) | 13 | 16 | 13 | 16
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 6 | 5 | 6
Hypertension (Vascular disorders) | 20 | 10 | 20 | 10
Phlebitis (Vascular disorders) | 6 | 7 | 6 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 7 | 6 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 5 | 4 | 5
Proteinuria (Renal and urinary disorders) | 6 | 5 | 6 | 5
Blood bilirubin increased (Investigations) | 1 | 3 | 0 | 5
Intestinal obstruction (Gastrointestinal disorders) | 1 | 3 | 2 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less